CLINICAL TRIAL: NCT02634658
Title: The Diagnosis and Incidence of Critical Illness Polyneuromyopathy in Medical and Neurosurgical ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-1557
Record Dates: First submitted 2015-11-13; First posted 2015-12-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — High-Energy Shock Waves; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical ICU Subjects (Experimental): All Medical ICU subjects that meet eligibility criteria and are enrolled in the study will receive muscle Ultrasounds, Nerve Conduction Studies and Electromyography (EMG).
  Interventions: Other: Muscle Ultrasound; Other: Nerve Conduction Study; Other: Electromyography
- Neuro ICU Subjects (Experimental): All Neuro ICU subjects that meet eligibility criteria and are enrolled in the study will receive Nerve Conduction Studies and Electromyography (EMG).
  Interventions: Other: Nerve Conduction Study; Other: Electromyography

INTERVENTIONS:
Other: Muscle Ultrasound — Ultrasound will be performed using a linear-array transducer with standardized gain and varying depth based on the amount of overlying soft tissue and muscle size. The subjects will be examined in the supine position with extended limbs and relaxed muscles. We will perform bilateral scans of the biceps, anterior forearm, and anterior thigh at standardized sites. For muscle echogenicity measurements, we will scan the same muscles at the same points.
  Other Names: US; Ultrasound
  Arms: Medical ICU Subjects
Other: Nerve Conduction Study — Nerve Conduction Studies will be performed using a Nicolet EDX using standard procedures. Repetitive stimulation of the median motor nerve are performed in all subjects. Bilateral sural, radial and median sensory nerves will be analyzed. We will only perform surface, not subdermal sensory recordings. The bilateral peroneal, tibial and median motor responses will be recorded over extensor digitorum brevis, abductor hallucis brevis, and abductor pollicis brevis muscles. The peroneal motor nerve will be stimulated at the fibular head and lateral popliteal fossa, recording from the tibialis anterior muscle. The compound motor action potential (CMAP) responses will be elicited from standard distal and proximal sites.
  Other Names: NCS
Other: Electromyography — EMG studies will be performed using standard precautions. Insertional activity, spontaneous activity, motor unit potential (MUP) morphology and recruitment/activation pattern will be recorded from some combination of the deltoid, triceps, biceps, first dorsal interosseous, abductor pollicis brevis, iliopsoas, vastus medialis, and tibialis anterior muscles. The specific muscles studied for each patient will vary according to the patient's level of consciousness and ability to activate the muscles either voluntarily or during spontaneous limb movement. If possible, we will try to examine 3 unilateral upper extremity and 3 unilateral lower extremity muscles. If a patient is not able to volitionally participate in EMG testing (by contracting their muscles on command), we will analyze insertional/spontaneous activity and potentially morphology/recruitment (e.g. stroking the sole of the foot to stimulate contraction of the tibialis anterior).
  Other Names: EMG

SUMMARY:
This study plans to learn more about whether simpler diagnostic tests can be used to identify the development of acute neuromuscular loss of function in patients with critical illness and respiratory failure receiving mechanical ventilation. ICU patients admitted to the University of Colorado Hospital will be screened for eligibility and enrollment in the study to receive weekly measurements of nerve and muscle function through nerve conduction studies (NCS), muscle ultrasound tests, and concentric needle electromyography (EMG) tests.

DETAILED DESCRIPTION:
This study plans to learn more about whether simpler diagnostic tests can be used to identify the development of acute neuromuscular loss of function in patients with critical illness and respiratory failure receiving mechanical ventilation. ICU patients admitted to the University of Colorado Hospital will be screened for eligibility and enrollment in the study to receive weekly measurements of nerve and muscle function through nerve conduction studies (NCS), muscle ultrasound tests, and concentric needle electromyography (EMG) tests.

Collected data includes the subject's age, gender, race, ethnicity, length of stay in ICU, time on mechanical ventilation and pertinent medical history that could indicate baseline neuromyopathy (CNS disease, diabetes, HIV, alcohol use disorder). Baseline neurological examination will be performed within 48 hours of meeting the inclusion criteria. This examination will include the level of consciousness, muscle tone, motor strength using the Medical Research Council (MRC) Scale, sensory function, muscle stretch reflexes, and plantar responses. For MRC testing, six muscle groups will be tested bilaterally: shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and foot dorsiflexion. Clinical weakness on examination (which is necessary to make the diagnosis of CIPNM (Critical Illness Polyneuropathy and Myopathy)) is defined as an MRC score equal to or less than 48 (maximum score is 60). If a subject cannot participate in any MRC strength testing (e.g. due to sedation or encephalopathy) they will be coded at the lowest level (most severe clinical weakness). Nerve conduction studies (NCS) and concentric needle electromyography (EMG) will be performed (as described below) on the same day as the initial neurological examination. The neurological examination and NCS/EMG will be repeated on a weekly basis until CIPNM is diagnosed or the subject is discharged from the ICU.

SPECIFIC AIM #1:

Aim 1.1: To determine whether amplitude reductions in the peroneal and sural nerve action potentials on NCS can serve as accurate screening tests for CIPNM in patients with acute respiratory failure.

Aim 1.2: To determine whether increased duration of the CMAP on NCS can serve as an accurate screening test for CIPNM in patients with acute respiratory failure.

Aim 1.3: To determine whether changes in muscle ultrasound echogenicity and/or thickness can serve as accurate screening tests for CIPNM in patients with acute respiratory failure.

Aim 1.4: To determine the incidence of CIPNM in patients with neurological critical illness (such as intraparenchymal and subarachnoid hemorrhage), which requires prolonged length of stay in a neurosurgical intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1.1-1.3, one of the following 2 sets of criteria are needed for inclusion

Set 1:

1. Acute respiratory failure defined as a Pa02 < 60 mm Hg on room air, the requirement of supplemental oxygen, or a PaC02 > 45 mm Hg.
2. Admission to an intensive care unit.
3. Mechanical ventilation support through an endotracheal tube for greater than 48 hours.
4. Severe sepsis (suspected or documented infection + at least 2/4 SIRS criteria + organ dysfunction) or septic shock (sepsis plus hypotension refractory to intravenous fluids or plasma lactate > 1.5 times the upper limit of normal)

Set 2:

1. Acute respiratory failure defined as requiring invasive or non-invasive ventilation with a p/f ratio ≤ 250
2. Admission to an intensive care unit, in ICU for greater than 48 hours.
3. Plus dysfunction in one of the following organ systems:

   1. Cardiovascular dysfunction: (at least one of the following) i. SBP ≤ 90 mm Hg or MAP ≤ 70 mm Hg for at least one hour despite adequate fluid resuscitation. Adequate fluid resuscitation is defined as the patient receiving intravenous fluid resuscitation of ≥ 30 mL/kg administered at any time during the 4 hours before a hypotensive blood pressure.

      ii. The use of vasopressors in an attempt to maintain a SBP of ≥ 90 mm Hg or a MAP of ≥ 65 mm Hg despite adequate intravascular volume status. Adequate intravascular volume status is defined as intravenous fluid resuscitation of ≥ 30 mL/kg administered at any time during the 4 hours before or after initiation of vasopressor therapy. Vasopressive therapy is defined as any one of the following: Norepinephrine, Phenylephrine, Epinephrine, Dopamine ≥ 5 mcg/kg/min, or Vasopressin ≥ 0.03 units/min.
   2. Kidney dysfunction: Urine output < 0.5 ml/kg of body weight/hr for 1 hour despite adequate fluid resuscitation or adequate intravascular volume status (as defined above)
   3. Hematologic dysfunction: Platelet count < 80,000 or a decrease by 50% over the previous 3 days.
   4. Acidosis: (at least one of the following) i. pH ≤ 7.30 ii. Plasma lactate > 1.5 times the upper limit of normal

For Aim 1.4, all of the following criteria are needed for inclusion.

1. Non-traumatic subarachnoid hemorrhage or intracerebral (intraparenchymal) hemorrhage.
2. Admission to a neurological or neurosurgical intensive care unit.
3. Mechanical ventilation support through an endotracheal tube for greater than 48 hours.

Exclusion Criteria:

For Aim 1.1-1.3:

1. Age less than 18 years.
2. Diagnosis of pre-existing disease of the peripheral motor or sensory nervous system or myopathy.
3. Central nervous system disorder that would compromise the ability of the patient to participate in the study.
4. Pharmacologic paralysis.
5. Absence of ability to test at least one arm and one leg with NCS/EMG (e.g. due to amputation or overlying equipment).
6. Decremental response on repetitive nerve stimulation.
7. External pacemaker wire.
8. Pregnancy.
9. Initiation of mechanical ventilation (invasive or non-invasive) and admission to the ICU both >120 hours (5 days) ago.
10. Referral from another hospital for patients that have required mechanical ventilation for more than 48 hours.
11. Inability to obtain informed consent or refusal to participate in the study.
12. Known steroid-induced myopathy prior to ICU admission resulting from chronic systemic glucocorticoid therapy.

For Aim 1.4:

1. Isolated subdural or epidural hematoma
2. Age less than 18 years.
3. Diagnosis of pre-existing disease of the peripheral motor or sensory nervous system or myopathy.
4. Pharmacologic paralysis.
5. Absence of ability to test at least one arm and one leg with NCS/EMG (e.g. due to amputation or overlying equipment).
6. Decremental response on repetitive nerve stimulation.
7. External pacemaker wire.
8. Pregnancy.
9. Initiation of mechanical ventilation and admission to the ICU both >120 hours (5 days) ago.
10. Referral from another hospital for patients that have required mechanical ventilation for more than 48 hours.
11. Inability to obtain informed consent or refusal to participate in the study. Known steroid-induced myopathy prior to ICU admission resulting from chronic systemic glucocorticoid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Aims 1.1-1.3: Number of medical ICU subjects diagnosed with CIPNM according to Moss/Quan established criteria of CIP or CIM. | Weekly up to Day 28 or hospital discharge whichever occurs first.
  Subjects have CIPNM if either Moss/Quan criteria for (CIP) or (CIM) criteria are met:
  CIP:
  SNAP amplitudes < 80% of lower norm limit of 2+ nerves, Reduced recruitment on EMG, Absence of decremental response, and MRC score < 48 or clinical weakness on exam
  CIM:
  SNAP amplitudes > 80% of the lower norm limit of 2+ nerves, CMAP amplitudes < 80% of the lower limit of normal in two or more nerves without conduction block, needle EMG with short-duration, low amplitude motor unit potentials with early recruitment, absence of a decremental response, and MRC score < 48 or clinical weakness on exam
  CIPNM:
  Absence of a decremental response, SNAP amplitudes < 80% of the lower limit of normal in two or more nerves, CMAP amplitudes < 80% of the lower limit of normal in two or more nerves without conduction block, sustained spontaneous activity and/or changes in motor unit recruitment, in at least two muscles, and MRC score < 48 or clinical weakness on exam
Aim 1.4: Number of neurosurgical ICU subjects diagnosed with CIPNM according to Moss/Quan established criteria of CIP or CIM. | Weekly through Day 28 or hospital discharge whichever occurs first
  Subjects have CIPNM if either Moss/Quan criteria for (CIP) or (CIM) criteria are met:
  CIP:
  SNAP amplitudes < 80% of lower norm limit of 2+ nerves, Reduced recruitment on EMG, Absence of decremental response, and MRC score < 48 or clinical weakness on exam
  CIM:
  SNAP amplitudes > 80% of the lower norm limit of 2+ nerves, CMAP amplitudes < 80% of the lower limit of normal in two or more nerves without conduction block, needle EMG with short-duration, low amplitude motor unit potentials with early recruitment, absence of a decremental response, and MRC score < 48 or clinical weakness on exam
  CIPNM:
  Absence of a decremental response, SNAP amplitudes < 80% of the lower limit of normal in two or more nerves, CMAP amplitudes < 80% of the lower limit of normal in two or more nerves without conduction block, sustained spontaneous activity and/or changes in motor unit recruitment, in at least two muscles, and MRC score < 48 or clinical weakness on exam

SECONDARY OUTCOMES:
ICU length of stay | upon completion of ICU stay, commonly 7-14 days.
  ICU length of stay
ICU-free days | upon completion of inpatient period, commonly up to 28 days.
  the number of days out of 28 that the subject is alive and out of the ICU, but remains hospitalized.
time on mechanical ventilation | upon completion of ventilation period, commonly 3-14 days.
  time on mechanical ventilation
hospital length of stay | upon completion of inpatient period, commonly up to 28 days.
  hospital total length of subject stay.
hospital-free days | 28 days
  the number of days oout of 28 that the subject was alive and out of the acute care hospital.
in hospital mortality | 28 days
  Incidence of in hospital mortality through day 28
Discharge location | up to 28 days
  Subject discharge location from acute hospitalization period to home, SNF, rehab hospital, LTACH, hospice, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided